CLINICAL TRIAL: NCT05401266
Title: The Effect of Mild Hypercapnia During Anesthetic Emergence on Recovery Time From TIVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-0389
Record Dates: First submitted 2022-05-26; First posted 2022-06-02 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-05

CONDITIONS: Total Intravenous Anesthesia
Keywords: hypercapnia; recovery time; total intravenous anesthesia
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal blood carbonic acid level (No Intervention): After propofol infusion was stopped, ventilation parameters were adjusted to maintain end-expiratory carbon dioxide (ETCO2) 35-40 mmHg until spontaneous respiration was restored.
- mild hypercapnia (Experimental): After propofol infusion was stopped, ventilation parameters were adjusted to achieve and maintain ETCO2 50-55 mmHg until spontaneous respiration was restored.
  Interventions: Procedure: mild hypercapnia

INTERVENTIONS:
Procedure: mild hypercapnia — Ventilation parameters were adjusted to achieve and maintain ETCO2 50-55 mmHg until spontaneous respiration was restored
  Arms: mild hypercapnia

SUMMARY:
We hypothesized that patients with mild hypercapnia during anesthetic emergence after TIVA had a shorter recovery time than patients with normal blood carbonate levels. We will select patients undergoing transurethral lithotripsy, who were expected to have mild postoperative pain, compare tracheal extubation time in patients with normal blood carbonic acid level and mild hypercapnia, to evaluate the effect of blood carbonic acid level during anesthetic emergence on recovery time from TIVA by. We also examined the changes of cerebral blood flow by TCD to investigate the possible mechanism of mild hypercapnia affecting the recovery time from TIVA.

DETAILED DESCRIPTION:
At present, there is no effective intervention method for the recovery of general anesthesia, and the elimination of anesthetic agents, especially from the brain is a decisive factor in the emergence from general anesthesia. Many studies have reported the effect of hypercapnia on recovery time from volatile anesthetics. Hypercapnia can increase cardiac output and cerebral blood flow, increasing the ability to remove volatile anesthetics from the brain and shortening the recovery time from anesthesia.

Propofol is becoming the most common intravenous agent used for induction as well as maintenance of total intravenous anesthesia (TIVA). Its rapid elimination from the blood and brain is expected to shorten the recovery time from TIVA. Only a few clinical studies have investigated the relationship between hypercapnia and emergence time with propofol anesthesia. But those studies may have been influenced by postoperative pain, so the recovery time cannot reflect propofol metabolism alone. Moreover, intraoperative hypercapnia may increase the need for intraoperative anesthetic agents by increasing the clearance of agents from the brain.

As a non-invasive method, Transcranial Doppler ultrasonography（TCD）can be used to monitor blood flow changes in different parts of cerebral arterial circle(Willis circle）, and its safety and effectiveness in perioperative related fields have been proved.

We hypothesized that patients with mild hypercapnia during anesthetic emergence after TIVA had a shorter recovery time than patients with normal blood carbonate levels. We will select patients undergoing transurethral lithotripsy, who were expected to have mild postoperative pain, compare tracheal extubation time in patients with normal blood carbonic acid level and mild hypercapnia, to evaluate the effect of blood carbonic acid level during anesthetic emergence on recovery time from TIVA by. We also examined the changes of cerebral blood flow by TCD to investigate the possible mechanism of mild hypercapnia affecting the recovery time from TIVA.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20-60 years, with American Society of Anesthesiology physical status 1 to 2, undergoing transurethral lithotripsy under TIVA with endotracheal intubation; voluntarily signed informed consent forms.

Exclusion Criteria:

* Patients with mental, pulmonary, cardiac, endocrine, neuromuscular, liver and nervous system diseases or a history of such diseases; Lung CT showed atelectasis, pulmonary infection and pleural effusion. Patients taking sedatives or other drugs that might interfere with the study; Alcohol or drug dependence; Patients who have had a history of general anesthesia within the past month; Patients with body mass index (BMI) of 30 kg/m2 or above; Patients who are expected to be under anesthesia for less than 30 minutes; Patients with difficult airways.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Tracheal extubation time | 1 year
  The time from propofol infusion stopped to Tracheal extubation

SECONDARY OUTCOMES:
Time of anesthesia | 1 year
  Time from anesthesia induction to cessation of propofol infusion
Total infusion of propofol and remifentanil | 1 year
  Total infusion of propofol and remifentanil
Spontaneous respiratory recovery time | 1 year
  The time from the beginning of cessation of propofol infusion to the time when the patient begins to cough or when the ETCO2 waveform changes
Time of eyes or mouth opening | 1 year
  The time from the beginning of cessation of propofol infusion to the time when patients can open their eyes or mouth
Changes in cerebral blood flow examined by transcranial Doppler (TCD) | 1 year
  Examine at the following four time points: before anesthesia induction; 10min after operation; After adjustment of ETCO2 is completed in post-anaesthesia care unit(PACU); 20 min after tracheal extubation

CONTACTS AND LOCATIONS:
Overall Officials: Li Li Fang, PhD, Study Director — Study Official Affiliation
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No